CLINICAL TRIAL: NCT06217432
Title: Tendinopathy: Optimal Time for Management Through Exercise (TENDOTIME) - a Randomised Controlled Study Comparing Targeted Training Performed Morning and Late Afternoon in a 12-week Intervention Program on Chronic Patellar Tendinopathy
Brief Title: A Study of the Effect of Time-of-day of Training on Chronic Patellar Tendinopathy
Acronym: TENDOTIME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Chloé Yeung, Senior Researcher, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: TENDOTIME
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Tendinopathy; Jumper's Knee
MeSH Terms: conditions — Tendinopathy | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Morning exercise (Experimental): Three sessions per week of targeted resistance exercise targeting the quadriceps muscles performed between 6:00 and 8:00 for 12 weeks.
  Interventions: Other: Resistance training for knee extensors
- Late afternoon exercise (Experimental): Three sessions per week of targeted resistance exercise targeting the quadriceps muscles performed between 16:00 and 18:00 for 12 weeks.
  Interventions: Other: Resistance training for knee extensors
- Healthy control (No Intervention): Healthy individuals without tendinopathy as controls for the transcriptomics and proteomics analyses.

INTERVENTIONS:
Other: Resistance training for knee extensors — The exercise will be started at 60% of 1 repetition maximum (RM) and progressed to 75% of 1 RM during the first 3 weeks and maintained throughout the intervention period. The exercise will be performed slowly (6 s/ repetition).
  Arms: Late afternoon exercise; Morning exercise

SUMMARY:
The study is a 12-week human study where 60 participants with chronic patellar tendinopathy (more than 3 months symptoms duration) are randomised to undergo 12 weeks of targeted resistance exercise either in the morning or in the late afternoon. The overall aim is to investigate when the best time of the day to perform muscular strength training therapy towards tendinopathy is. The study will also include 10 healthy controls who will not perform any exercise training.

ELIGIBILITY:
Inclusion Criteria:

* Sports active men and women
* Age (18-55) years old
* BMI (18.5-30)
* Uni- or bilateral patellar tendinopathy
* Symptom onset >90 days ago

Exclusion Criteria:

* Patellar tendinopathy longer than 24 months
* Previous surgery in the knee on the ipsilateral side
* Corticosteroid injection in the patellar tendon on the ipsilateral side within the last 6 months
* Any confounding diagnosis to the knee joint
* Known arthritis
* Known diabetes
* Known rheumatic disorders
* Inability to follow rehabilitation or complete follow-ups
* Enrolled in a resistance based-rehabilitation program for the affected patellar tendon within the previous 3 months
* Have an occupation where it is not feasible to avoid pain provoking tasks
* Pregnancy
* Have sleeping disorders or disruptions, e.g., night shift work
* Use of medicines or supplements known to affect collagen synthesis or sleep

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Patient perception VISA-P | Change from baseline at week 12.
  Change in Victorian Institute of Sports Assessment - patella (VISA-P) total score. The VISA-P asses symptoms, function and the ability to participate in sport. It consists of 8 questions, with a maximum score of 100 indicating the person is asymptomatic and fully per-forming and lower scores indicating more symptoms and limitations of function and activity.

SECONDARY OUTCOMES:
Patient perception VISA-P truncated | Change from baseline at week 12 and 52.
  Change in Victorian Institute of Sports Assessment - patella (VISA-P) truncated score. The truncated score only including questions 2-6, with a maximum score of 50. Lower scores indicating more symptoms and limitations of function and activity.
Patient perception VISA-P | Change from baseline at week 52.
  Change in Victorian Institute of Sports Assessment - patella (VISA-P) total score. The VISA-P asses symptoms, function and the ability to participate in sport. It consists of 8 questions, with a maximum score of 100 indicating the person is asymptomatic and fully per-forming and lower scores indicating more symptoms and limitations of function and activity.
Self-reported improvement (GROC) | Change from baseline at week 12 and 52.
  Self-reported improvement after treatment will be evaluated by the Global Rating of change (GROC) on a 7-point Likert scale ranging from 'much improved' to 'much worse'.
Self-reported satisfaction (PASS) | Change from baseline at week 12 and 52.
  Self-evaluated satisfaction with treatment result will be evaluated by Patient Acceptable Symptom State (PASS) on a 5-point Likert scale ranging from 'very satisfied' to 'very unsatisfied'.
Counter movement jump height | Change from baseline at week 52.
  Jump height during counter movement jump test will be used to assess patellar tendinopathy caused functional deficits.
Pain during single-leg decline squat (SLDS) | Change from baseline at week 12 and 52.
  Participants performed a decline squat on a 25°decline board and reported pain using an 11 point numeric rating scale (NRS) upon completion, with 10 being the worst imaginable pain and 0 denoting no pain.
Ultrasonography - tendon thickness | Change from baseline at week 12 and 52.
  Grey scale ultrasonography will be used for evaluation of patellar tendon thickness.
Ultrasonography - power Doppler | Change from baseline at week 12 and 52.
  Doppler ultrasonography will be used for evaluation of patellar tendon vascularization/blood flow.
Lean mass by dual-energy X-ray absorptiometry | Change from baseline at week 12.
  Change in quadriceps lean muscle mass by DEXA.
Expression of circadian clock genes | Change from baseline at week 12, compared to healthy controls.
  Changes in expression of circadian clock genes and known tendon clock target genes by tendon tissue biopsies measured in the bulk RNA by RNA sequencing and reverse transcription-quantitative polymerase chain reaction (RT-qPCR).
Expression of extracellular matrix (ECM) and ECM regulator genes | Change from baseline at week 12, compared to healthy controls.
  Changes in expression of ECM and ECM regulator genes by tendon tissue biopsies measured in the bulk RNA by RNA sequencing and reverse transcription-quantitative polymerase chain reaction (RT-qPCR).
Global expression of genes | Change from baseline at week 12, compared to healthy controls.
  Unbiased examination of global changes in expression of genes by tendon tissue biopsies measured in the bulk RNA by RNA sequencing.
Histochemical staining of tendon sections | Change from baseline at week 12, compared to healthy controls.
  Morphology of tendon tissue regions, including cells and blood vessels, measured by histochemical and immunohistochemical stainings of tendon tissue biopsies.
Spatial changes of gene expression | Change from baseline at week 12, compared to healthy controls.
  Unbiased examination of global changes in expression of genes in regions of interests of tendon tissue biopsies measured by spatial transcriptomics.
Spatial changes of extracellular matrix protein levels | Change from baseline at week 12, compared to healthy controls.
  Unbiased examination of global changes in levels of extracellular matrix proteins in regions of interests of tendon tissue biopsies measured by spatial transcriptomics.
Blood samples | Change from baseline at week 12, compared to healthy controls.
  Identification of potential biomarkers of tendon injury and repair by metabolomics and proteomics.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sports Medicine Copenhagen, Copenhagen NV, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Undecided